CLINICAL TRIAL: NCT06732856
Title: A Phase Ib/II Trial of Neoadjuvant Zolbetuximab Plus Docetaxel, Oxaliplatin and S-1 Chemotherapy in Patients With Locally Advanced Gastric Cancer
Acronym: NEO-CLAUD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2402
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stomach Neoplasm; Gastric (Stomach) Cancer
Keywords: NEO-ADJUVANT; ADJUVANT; distant metastasis limited to lymph node gastric cancer; unresectable locally advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — zolbetuximab; Oxaliplatin; Docetaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: zolbetuximab; Drug: Oxaliplatin; Drug: Docetaxel; Drug: S-1

INTERVENTIONS:
Drug: zolbetuximab — 1. Neoadjuvant treatment
     : Zolbetuximab 800*/600 mg/m2 Q3W on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles.
     (*Loading dose of zolbetuximab (800 mg/m²) on C1D1, followed by subsequent doses of 600 mg/m² every 3 weeks)
  2. Surgery
     : Total gastrectomy (TG) or distal gastrectomy (DG) accompanied with dissection of the D2 lymph node
  3. Adjuvant treatment After 3-8 weeks from surgery, S-1 40/50/60 mg/m2 bid orally on D1-28 plus Zolbetuximab 600 mg/m2 on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.
Drug: Oxaliplatin — 1. Neoadjuvant treatment : Zolbetuximab 800*/600 mg/m2 Q3W on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles. (*Loading dose of zolbetuximab (800 mg/m²) on C1D1, followed by subsequent doses of 600 mg/m² every 3 weeks) 2. Surgery : Total gastrectomy (TG) or distal gastrectomy (DG) accompanied with dissection of the D2 lymph node 3. Adjuvant treatment After 3-8 weeks from surgery, S-1 40/50/60 mg/m2 bid orally on D1-28 plus Zolbetuximab 600 mg/m2 on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.
Drug: Docetaxel — 1. Neoadjuvant treatment : Zolbetuximab 800*/600 mg/m2 Q3W on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles. (*Loading dose of zolbetuximab (800 mg/m²) on C1D1, followed by subsequent doses of 600 mg/m² every 3 weeks) 2. Surgery : Total gastrectomy (TG) or distal gastrectomy (DG) accompanied with dissection of the D2 lymph node 3. Adjuvant treatment After 3-8 weeks from surgery, S-1 40/50/60 mg/m2 bid orally on D1-28 plus Zolbetuximab 600 mg/m2 on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.
Drug: S-1 — 1. Neoadjuvant treatment : Zolbetuximab 800*/600 mg/m2 Q3W on day (D) 1, Docetaxel 50 mg/m2 intravenously (IV) on D1, oxaliplatin 100 mg/m2 IV on D1, S-1 40 mg/m2 bid orally on D1-14, will be administered every three weeks for three cycles. (*Loading dose of zolbetuximab (800 mg/m²) on C1D1, followed by subsequent doses of 600 mg/m² every 3 weeks) 2. Surgery : Total gastrectomy (TG) or distal gastrectomy (DG) accompanied with dissection of the D2 lymph node 3. Adjuvant treatment After 3-8 weeks from surgery, S-1 40/50/60 mg/m2 bid orally on D1-28 plus Zolbetuximab 600 mg/m2 on D1 and D22 will be administered every 6 weeks for 12 months as an adjuvant treatment.

SUMMARY:
Claudin 18.2 is a promising therapeutic target overexpressed on the surface of gastric cancer cells. The addition of zolbetuximab, the monoclonal antibody targeting Claudin 18.2 to chemotherapy in two recent Phase 3 studies prolonged survival outcomes, indicating that Claudin 18.2 is a valid target in gastric cancer. Asan Medical Center researchers conducted a study on Claudin 18.2 expression in patients with operable gastric cancer and defined moderate to strong claudin expression in more than 75% of tumor cells as Claudin 18.2 overexpression, which was observed in 46.5% of patients with stage I-III tumors. This suggests that zolbetuximab-based treatment may be possible in patients with LAGC.

Therefore, The investigator designed a prospective, multicenter, open-label, Phase Ib/II study to determine the efficacy and safety of zolbetuximab/DOS as neoadjuvant chemotherapy in patients with LAGC.

DETAILED DESCRIPTION:
Although the global incidence and mortality of gastric cancer has declined in recent decades, gastric cancer is the fifth most common cancer and the third leading cause of cancer-related death. Surgical resection is the main treatment for patients with localized gastric cancer. However, postoperative recurrences are common, and approximately 40% of patients experience recurrences 2 years after surgery.

Various adjuvant therapies have been studied over the past decades to improve the rate of postoperative recurrences. Perioperative chemotherapy and postoperative chemoradiotherapy or adjuvant chemotherapy has been shown to improve overall survival in patients with resectable gastric cancer. The preferred treatment strategy is chosen according to the expected locoregional control after surgery, and tends to vary depending on the geographical location.

Two large randomized, controlled, Phase 3 trials in East Asia investigated the efficacy of S-1 for 1 year or capecitabine and oxaliplatin (XELOX) for 6 months as adjuvant chemotherapy following D2 gastrectomy compared to D2 gastrectomy alone in patients with resectable gastric cancer. Both studies showed an apparent benefit of adjuvant chemotherapy versus surgery alone in survival, with 5-year overall survival rates of 70 to 80% in patients receiving adjuvant chemotherapy and 60 to 70% in patients receiving surgery alone. Based on these results, D2 gastrectomy with S-1 or XELOX as adjuvant chemotherapy is the treatment strategy generally selected for patients with resectable gastric cancer in East Asia. However, approximately 30 to 35% of patients experience disease recurrence despite the addition of adjuvant chemotherapy, suggesting that a better treatment strategy needs to be developed in this clinical setting.

One of the strategies for improving survival outcomes of locally advanced gastric cancer may be the introduction of neoadjuvant chemotherapy. Recently, the pivotal phase 3 PRODIGY and RESOLVE studies have demonstrated survival benefits of adding neoadjuvant chemotherapy to surgery followed by adjuvant chemotherapy over up-front surgery followed by adjuvant chemotherapy in Asian patients. Based on these results, neoadjuvant chemotherapy is considered one of the viable options for patients with locally advanced gastric cancer.

Claudin 18.2 is a promising therapeutic target overexpressed on the surface of gastric cancer cells. The addition of zolbetuximab, the monoclonal antibody targeting Claudin 18.2 to chemotherapy in two recent Phase 3 studies prolonged survival outcomes, indicating that Claudin 18.2 is a valid target in gastric cancer. Asan Medical Center researchers conducted a study on Claudin 18.2 expression in patients with operable gastric cancer and defined moderate to strong claudin expression in more than 75% of tumor cells as Claudin 18.2 overexpression, which was observed in 46.5% of patients with stage I-III tumors. This suggests that zolbetuximab-based treatment may be possible in patients with LAGC.

Therefore, the investigator designed a prospective, multicenter, open-label, Phase Ib/II study to determine the efficacy and safety of zolbetuximab/DOS as neoadjuvant chemotherapy in patients with LAGC.

< Primary objective(s)>

* RP2D (phase Ib part)
* Pathologic complete regression rate (pCR) (phase II part)

< Secondary objective(s)>

* Progression-free survival by RECIST v1.1
* Overall survival (OS)
* Overall response rate (ORR) during by RECIST v 1.1
* Disease control rate (DCR) by RECIST v 1.1
* Safety profiles by

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, pathologically confirmed, potentially resectable gastric or gastroesophageal junction adenocarcinoma
2. Subjects who are CLDN18.2 positive (VENTANA 43-14A ≥75%)
3. Patients with clinical stage T3-4/N0 or T2-4/N+ on CT according to the American Joint Committee on Cancer (AJCC) 8th edition
4. If suspected by CT, patient who has not been confirmed to have peritoneal seeding by laparoscopy
5. Subject able to provide signed informed consent form, including compliance with the requirements and contraindications specified in the informed consent form (ICF) and in this protocol
6. Patients aged 19 years or older at study entry
7. Patient with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
8. Patient with expected survival >12 months
9. Weight >30 kg
10. Patient without neuropathy A. Grade 1 is allowed based on NCI CTCAE v5.0. B. Grade 2 or higher is excluded based on NCI CTCAE v5.0
11. Individual with confirmed adequate normal organ and bone marrow function, as defined in the applicable items below:

    * Hemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) >1.5 x 103/mcL (>1,500 per mm3)
    * Platelet count ≥100 x 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional ULN
    * Measured creatinine clearance (CL) >40 mL/min or creatinine CL >40 mL/min as calculated by Cockcroft-Gault formula (Cockcroft and Gault 1976) or based on a 24-hour urine sample for determination of creatinine clearance

      1. Male creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x Serum creatinine (mg/dL)
      2. Female creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x Serum creatinine (mg/dL) x 0.85
12. Evidence of menopause, or negative urine/blood pregnancy test in premenopausal women; women with amenorrhea for at least 12 months without any other medical cause are considered menopausal. The following age requirements apply:

    * A woman under age 50 is considered menopausal if 1) she has had amenorrhea for at least 12 months without hormone therapy, and 2) her LH and FSH blood levels are at menopausal levels or she has undergone bilateral oophorectomy, hysterectomy, etc.
    * A woman aged 50 years or older is considered menopausal if

      1. she has had amenorrhea for at least 12 months without hormone therapy, or
      2. she became menopause after 1 year of amenorrhea following radiation or anticancer treatment, or
      3. she has undergone bilateral oophorectomy, bilateral salpingectomy, hysterectomy, etc.
13. Patient who is willing and able to comply with the protocol during the study, including treatments and tests such as scheduled visits, follow-up, etc.

Exclusion Criteria:

1. Patient who received investigational product in another clinical study 2 weeks prior to participation in this clinical study
2. Patient currently enrolled in another clinical study, other than the observational (non-interventional) study or follow-up period of an interventional clinical study.
3. Concomitant chemotherapy, immunotherapy, biologic or hormonal therapy. Hormonal therapies not related to treatment for cancer (e.g., hormone replacement therapy) are allowed.
4. Major surgical procedure within 28 days prior to zolbetuximab administration
5. Distant metastasis including M1 lymph node
6. Patient unable to take oral medication
7. Gastric outlet obstruction and/or severe gastrointestinal hemorrhage that restricts diet without treatment
8. Impaired intestinal absorption, including:

   * Intestinal obstruction
   * Chronic inflammatory bowel disease
   * Operation history of extended bowel resection
   * Gastric dumping syndrome
9. Patient with a history of organ transplant
10. Uncontrolled intercurrent disease including, but not limited to:

    Ongoing or active infection, congestive heart failure with symptoms, uncontrolled hypertension, unstable angina, arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions accompanied with diarrhea, mental illness or social conditions that prevent compliance with study requirements, significantly increase the risk of adverse reactions, or interfere with written consent
11. History of other primary malignancy, with the exception of:

    * Patient who is at low risk of recurrence with disease-free status for at least 5 years prior to starting chemotherapy due to curative treatment
    * Patient who is currently disease-free with cured skin cancer (except melanoma) or lentigo maligna
    * Patient who is currently disease-free with cured in situ carcinoma
12. Patient with a history of active congenital immunodeficiency
13. Active infection, such as tuberculosis, confirmed by history, physical examination, radiographic findings, and TB testing per local standards, or HIV.

    * Tuberculosis: History, physical examination, or radiological findings suggestive of active tuberculosis, or tuberculosis confirmed by tuberculosis testing per local standards (active TB is excluded and old TB is allowed)
    * For HBV infection, the patient may be enrolled if appropriately treated with antiviral agents, etc.
    * HIV

      1. HIV Ag/Ab: If reactive, exclude
      2. HIV Ag/Ab: If non-reactive, enroll
14. Pregnant or lactating woman and man or woman of childbearing potential who is unwilling to use effective contraception (from the screening period to 90 days after the last dose of zolbetuximab)
15. Individual with known allergy and hypersensitivity to the investigational product or its components

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of R0 resection rate in patients who underwent prior chemotherapy as a clinical trial.(phase II part) | 1 year
  Evaluation of R0 resection rate.
Recommended phase 2 dose (RP2D) (phase Ib part) | 1 year
  Recommended phase 2 dose (RP2D) (phase Ib part)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea